CLINICAL TRIAL: NCT01880411
Title: Phase I, Open-Label Study of the Safety, Tolerability, and Immunogenicity of a Three Dose Regimen of Escalating Doses of PEK Fusion Protein Vaccine (PEK + GPI-0100) in Patients With LSIL or HSIL
Brief Title: Phase I, Open-Label Study of the Safety, Tolerability, and Immunogenicity PEK Fusion Protein Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HealthBanks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBPEKVPI001
Record Dates: First submitted 2013-06-13; First posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: PEK fusion protein Healthbanks
MeSH Terms: conditions — Uterine Cervical Dysplasia

ARMS (1):
- PEK Fusion Protein Vaccine (Experimental): PEK Fusion Protein Vaccine Injection 0.1mg, 0.3mg and 1.2mg One injection at one week intervals
  Interventions: Biological: PEK Fusion Protein Vaccine

INTERVENTIONS:
Biological: PEK Fusion Protein Vaccine — PEK (PE-E7-K3), a recombinant protein combined with GPI-0100 adjuvant

SUMMARY:
Phase I, Open-Label Study of the Safety, Tolerability, and Immunogenicity of a Three Dose Regimen of Escalating Doses of PEK Fusion Protein Vaccine in Women with LSIL or HSIL.

PEK fusion protein vaccine (PEK + GPI-0100) is safe and well tolerated in patients with low-grade squamous intraepithelial lesions (LSIL) or high grade squamous intraepithelial lesions (HSIL) of the cervix and induces a measurable immune response.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18 to 45 years
* Written informed consent in accordance with institutional guidelines
* Negative pregnancy test
* LSIL or HSIL on Papanicolaou (PAP) smear within the prior 6-8 weeks
* Normal electrocardiogram (ECG), laboratory values (chemistry, complete blood count) and urinalysis, as judged by Grade 0-1 as per National Cancer Institute Common Toxicity Criteria (NCI-CTC) performed up to 30 days prior to administration of study treatment.
* Body mass index (BMI) ≤32 kg/m2
* Women of child-bearing potential (WOCBP) agree to use two forms of medically effective contraception (e.g. hormonal contraception, intrauterine device, barrier method, spermicide, etc…) during the study and for at least 12 weeks following the completion of treatment. Patients agree to inform the investigator immediately if they become pregnant during the study or within 12 weeks following completion of treatment and to provide information about the pregnancy, delivery and health of the infant until the age of one month.
* Able and willing to comply with all study procedures

Exclusion Criteria:

* Active infection with herpes simplex virus (HSV)
* Positive serologic test for human immunodeficiency virus (HIV), Hepatitis C virus (HCV), or Hepatitis B surface antigen (HBsa)
* Pregnant or breast-feeding
* History of any prior cervical surgical treatment
* History of any active autoimmune disease or current medical condition requiring the use of systemic or topical corticosteroids (excluding steroid containing eye drops or inhaled steroids) or other immunosuppressive agents within 4 weeks prior to enrollment
* History of cancer (excluding basal cell carcinoma of the skin)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Administration of any blood product within 3 months of enrollment
* Administration of any vaccine within 6 weeks of enrollment
* Active infection requiring antimicrobial treatment
* Participation in any study with an investigational compound or device within 30 days prior to signing informed consent
* Any hematologic disorder involving platelets or clotting abnormalities or any condition requiring treatment with transfusions, anticoagulants or platelet inhibitors
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study protocol
* Any condition which, in the opinion of the investigator, would limit the evaluation of the patient.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Christina S Chu, MD, Principal Investigator — University of Pennsylvania